CLINICAL TRIAL: NCT06391658
Title: Eight Weeks of Functional Training Improves the Functional Capacity and Physical Fitness of People Whit Spinal Cord Injury After Social Distancing Due to the Covid-19 Pandemic
Brief Title: Functional Training Improves the Functional Capacity and Physical Fitness of People Whit Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 54458021.8.0000.5235
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Physical Exercise; Disability Physical
Keywords: Rehabilitation; Spinal Cord Injury; Physical Disability; Physical Training.COVID-19
MeSH Terms: conditions — Motor Activity; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FT group (Experimental): Functional Training group
  Interventions: Other: Functional Training

INTERVENTIONS:
Other: Functional Training — Functional training was performed for eigth weeks. The group participated on the supervised training once a week and twice a week at home. The training was arranged in a circuit method, consisting of three to four blocks with two to three exercises each, with an execution time of two minutes and recovery of thirty seconds between exercises and one minute between each block. The exercises emphasized integrated, functional and multi-joint movements for mobility, flexibility, strength, power and muscular endurance with overload, as well as agility, speed and balance exercises.

SUMMARY:
The aim of this study is to understand the effect of adapted functional training on the physical fitness, functionality and quality of life of individuals with SCI after social distancing due to COVID-19. The main question[s] it aims to answer are:

* Are the participants of the functional training program adapted for people with spinal cord injury show better results in functional capacity in post-test evaluations training period, when compared to your results in the functional training pré-period?
* Is adapted functional training capable of improving cardiorespiratory fitness, muscular strength and body composition?
* Can the perception of quality of life be influenced by functional training?

Participants will be evaluated through questionnaires and field tests, such as:

* Functional Capacity (battery of motor tests related to functional independence and Motor Assessment Scale),
* Physical fitness (handgrip test; medicine ball throw; Illinois agility and 12-minute displacement) and Quality of Life (WHOQOL-DIS).

DETAILED DESCRIPTION:
The spinal cord is an important component of the central nervous system, whose function is to transmit motor nerve impulses from the brain to other parts of the body, and to transmit sensory impulses from other systems of the body to the brain. Among adults living with SCI, studies show that participation in physical exercise programs, such as functional training, is associated with numerous health-related benefits, including improvements in cardiorespiratory fitness, energy production, and muscle strength, reduced the risk of cardiometabolic diseases and osteoporosis, in addition to psychosocial and quality of life benefits. However, high rates of physical inactivity among people with SCI are still a reality and, therefore, a cause for medical and health concern. In the recent scenario, measures to prevent and contain COVID-19 further contributed to the increase in sedentary time and behavior among individuals with spinal cord injury. Considering that TF aims to enhance specific actions in activities of daily living, the hypothesis of the cohort study is that a positive effect will be observed on functional capacity, on elements of physical fitness of these individuals and on quality of life after 8 weeks of training functional. Participants will be recruited by convenience and will undergo assessments of body composition, functional capacity, physical fitness and quality of life pre and post eight weeks of functional training, three times a week.

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* Aged 18 or over
* Have had Spinal Cord Injury for at least two years
* Wheelchair users

Exclusion Criteria:

* Individuals who had clinical or physical conditions that prevented them from carrying out the proposed tests

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Functional capacity with Battery of Motor Tests related to Functional Independence | Eigth weeks
  The Motor Test Battery consisted of function and reach tests. After adding up the test scores, the individuals were classified as: "complete dependence" (0 to 6 points), "moderate autonomy" (7 to 13 points), "high autonomy" (14 to 20 points) and "total autonomy" (21 to 27 points).
Functional capacity with Motor Assessment Scale | Eigth weeks
  The Motor Assessment Scale (Jorgensen et al., 2011) consists of six tests to assess static and proactive balance control, with the starting position being sitting on a bench, with hips and knees at 90º, without back support and feet on the floor. In each test, the testee can receive a score of 0 (does not perform the task and disqualifies the individual) or 1 (performs the task), with three possible attempts each.
Isometric handgrip strength | Eigth weeks
  To assess physical fitness through musculoskeletal capacity, the Lafayette hand dynamometer hand grip test (kgf; Lafayette hand dynamometer; United States) was used in three attempts for both sides, where the highest number achieved was validated, with the measurements measured in KGF.
Upper limb power | Eigth weeks
  A 3kg medicine ball throw test was carried out to assess the participant's muscle power. The participant had three attempts to throw the medicine ball as far as possible, with both hands at chest height. The distance, in meters (m), between the point where the ball touched the ground and the participant was measured and the lowest result of the three attempts was validated.
Agility | Eigth weeks
  The Illinois Agility Test was carried out, which is used to measure multidirectional agility, both for disabled people in wheelchairs and for non-disabled people in clinical or athletic situations. To carry out the test, cones were used to mark out a pre-established route to be covered in the shortest time possible. The participant could make three attempts and the one with the shortest time, measured in seconds (s), was validated.
Aerobic capacity | Eigth weeks
  Cardiorespiratory capacity was measured using the 12-minute walk test on a pre-defined course that was 25 meters long, 15 meters wide and marked off 2 meters at the corners, giving a total perimeter of 75.32 meters. The participants were asked to cover as much distance as possible, measured in miles (mi), during the 12 minutes.

SECONDARY OUTCOMES:
Arm muscle circumference | Eigth weeks
  Arm muscle circumference was calculated using the equations proposed by Gurney and Jelliffe (1973): CMB (cm) = [Arm circumference (cm) - (π x triceps skinfold (mm))]
Perceived quality of life | Eigth weeks
  Quality of life was investigated by applying the World Health Organization Quality of Life Questionnaire for People with Disabilities module ((WHOQOL-DIS), in the version translated and validated for Portuguese (Bredemeier et al., 2014). The options for each item are described on a five-level Likert scale, where participants rate satisfaction from 1 to 5 (5 "totally agree" and 1 "totally disagree"). The results were presented on a scale of 0 to 100 (WHOQOL,1998), scaled in a positive direction. In other words, the higher the score, the greater the interviewee's perception of QoL in each domain (WHOQOL,1998).

OTHER OUTCOMES:
Total body mass | Eigth weeks
  The measurement of total body mass was carried out with the participant in his wheelchair, using a scale of adequate dimensions, with an accuracy of 0.1 kg (ID-M300/5, Filizola, Brazil) and measurement unit in kilogram (kg). To determine the final TBM, the weight of the wheelchair was discounted.
Height | Eigth weeks
  Height was measured with the participant in a supine position on a stretcher (tape measure with a precision of 0.1 cm; CESCORF, Brazil) and measured in centimeters (cm). Height in dorsal decubitus was measured as the distance between the plane of the vertex and the calcaneus.
Body perimeters | Eigth weeks
  The body perimeters of the relaxed and contracted arm and the abdomen were measured. A tape measure with a precision of 0.1 cm was used (Cescorf, Brazil).
Triceps skinfold | Eigth weeks
  The triceps skinfold was measured with a 0.1 mm calibrated plicometer (Cescorf, Brazil)
Maximum oxygen consumption | Eigth weeks
  Based on the distance achieved, maximum oxygen consumption (VO2max) was estimated using the formula proposed by Franklin et al. (1990): VO2max (ml/kg/min) = (Distance miles - 0.37) /0.0337.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Barranco, Principal Investigator — Centro Universitário Augusto Motta
Locations (1):
- Centro Universitário Augusto Motta, Rio de Janeiro, Brazil